CLINICAL TRIAL: NCT00798109
Title: An Open Multicentric Randomized Clinical Trial Assessing the Impact of Motivational Interviewing on Cannabis Consumption in Patients With Psychiatric Disease
Brief Title: Effect of Motivational Therapy on Schizophrenia With Cannabis Misuse
Acronym: SCHIZOCAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 070156; AOM 07007 (Other: French Ministry)
Record Dates: First submitted 2008-09-30; First posted 2008-11-25 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Cannabis Dependence, Continuous
Keywords: Schizophrenia; Cannabis misuse comorbidity; Motivational interview; Randomised open trial
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Therapy (Experimental): Four motivational interview for cannabis abuse in schizophrenia population during one month
  Interventions: Behavioral: Motivational therapy
- Usual Care (Other): Usual care with intensive psychotherapy
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Motivational therapy — One hour of motivational therapy each weak during 4 weeks
  Arms: Motivational Therapy
Behavioral: Usual care — Patients received at least six hour of usual therapy, as in the experimental group
  Arms: Usual Care

SUMMARY:
Schizophrenia is a severe mental illness with a lifetime morbidity risk close to 1 %, involving both genetic and environmental risk factors. Prospective studies have shown that heavy use of cannabis in adolescence moderately increases the risk of developing schizophrenia. Many data have also suggested that the co-occurrence of cannabis abuse in patients with schizophrenia has a deleterious impact on the clinical outcome of schizophrenia. Cannabis abuse by schizophrenic patients is a significant public health problem for which there is no empirically validated treatment. We are presently studying the efficiency of motivational therapy on cannabis consumption in patients with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness with a lifetime morbidity risk close to 1 %, involving both genetic and environmental risk factors. Prospective studies have shown that heavy use of cannabis in adolescence moderately increases the risk of developing schizophrenia. Many data have also suggested that the co-occurrence of cannabis abuse in patients with schizophrenia has a deleterious impact on the clinical outcome of schizophrenia. Cannabis abuse by schizophrenic patients is a significant public health problem for which there is no empirically validated treatment. We are presently studying the efficiency of motivational therapy on cannabis consumption in patients with schizophrenia.

330 patients with schizophrenia and cannabis abuse or dependence (according to DSM-IV criteria) are randomly assigned to 4 motivational interview during one month or usual intensive treatment. Treatment is conducted in outpatient which are evaluated at the inclusion and at 6 month with Time-Line Follow Bach for the consumption, PANSS score, number of relapse…). A outcome measure was urinalysis results providing an objective measure of cannabis use throughout the six month of the trial.

ELIGIBILITY:
INCLUSION CRITERIA:

* Schizophrenia or schizo-affective disorder according to DSM-IV criteria
* Meeting DSM-IV criteria for actual cannabis abuse or dependance
* in current and regular contact with mental health service
* with an age at interview of 18 years or more
* No evidence of organic brain disease or clinically significant concurrent medical illness or learning disability
* Written informed consent was obtained from all subjects (patients and parents).

EXCLUSION CRITERIA:

* Not membership to a regime of social security or to a CMU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-11; Primary Completion 2012-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cannabis consumption evaluated by the Time-Line Follow Back at 6 months with mean percentage of abstinent day | inclusion, 3 month, 6 month, 12 month

SECONDARY OUTCOMES:
PANSS, GAF, number of DSM-IV criteria of cannabis dependence, May scale for treatment response, SF-12, la URICA, number of hospitalisation, mean number of joints per week, D9THC urinanalysis at 6M and cannabis consumption evaluated by the TLFB at 6M | inclusion, 3 month, 6 month, 12 month. Only inclusion and 6 month for urianalysis
  PANSS : global, positive, negative, general scores

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DUBERTRET, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de psychiatrie (Pr Adès), Colombes, France